CLINICAL TRIAL: NCT03833440
Title: Precision Immuno-Oncology for Advanced Non-small Cell Lung Cancer Patients With PD-1 ICI Resistance (PIONeeR Clinical Study)
Brief Title: Precision Immuno-Oncology for Advanced Non-small Cell Lung Cancer Patients With PD-1 ICI Resistance
Acronym: PIONeeR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-21; 2018-000914-39 (EudraCT Number)
Record Dates: First submitted 2019-02-05; First posted 2019-02-07 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; monalizumab; ceralasertib; Docetaxel; 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine

STUDY DESIGN:
Intervention Model Description: Arm A: combination of Durvalumab + NKG2A inhibitor Monalizumab (IPH2201), to target a PD-L1 co-inhibitory pathway
  * Arm B: combination of Durvalumab + CD73 antibody MEDI9447, to target limitations of antitumor T-cell immunity caused by adenosine receptor signaling
  * Arm C: combination of Durvalumab + ATR inhibitor AZD6738, to potentially enhance anti- tumour T-cell responses
  * Arm D: a standard third or forth-line chemotherapy maintenance (Docetaxel).
  * Arm E : combination of Durvalumab + MET kinase inhibitor Savolitinib (AZD6094)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Durvalumab + Monalizumab (Experimental)
  Interventions: Drug: Durvalumab (MEDI4736); Drug: Monalizumab (IPH2201)
- Durvalumab + MEDI9447 (Experimental)
  Interventions: Drug: Durvalumab (MEDI4736); Drug: Oleclumab (MEDI9447)
- Durvalumab + AZD6738 (Experimental)
  Interventions: Drug: Durvalumab (MEDI4736); Drug: Ceralasertib (AZD6738)
- Docetaxel (Active Comparator)
  Interventions: Drug: DOCETAXEL
- durvalumab+savolitinib (Experimental)
  Interventions: Drug: Durvalumab (MEDI4736); Drug: Savolitinib

INTERVENTIONS:
Drug: Durvalumab (MEDI4736) — 1500 mg, every 4 weeks. CxD1 for each cycle, 1 cycle = 28 days
  EXCEPT FOR CYCLE 1 IN ARM C : at C1D8 and cycle 1 = 35 days
  c=cycle D= day
  Arms: Durvalumab + AZD6738; Durvalumab + MEDI9447; Durvalumab + Monalizumab; durvalumab+savolitinib
Drug: Monalizumab (IPH2201) — 1500 mg, every 4 weeks. CXD1 for each cycle, 1 cycle = 28 days
  c=cycle D= day
  Arms: Durvalumab + Monalizumab
Drug: Oleclumab (MEDI9447) — 3000 mg every 2 week x 4 doses, followed by 3000 mg every 4 weeks. C1D1, C1D15, C2D1, C2D15 and CXD1 for the orther cycles, 1 cycle = 28 days.
  c=cycle D= day
  Arms: Durvalumab + MEDI9447
Drug: Ceralasertib (AZD6738) — 240 mg bid in Cycle 1, Days 1-7, followed by 7 days on treatment in each cycle between Days 22 and 28.
  CxD22-D28 for each cycle, 1 cycle = 28 days EXCEPT FOR CYCLE 1 : at C1D1,C1D29 and cycle 1 = 35 days
  c=cycle D= day
  Arms: Durvalumab + AZD6738
Drug: DOCETAXEL — 75 mg/m2, every 3 weeks. CxD1 for each cycle, 1 cycle = 21 days
  c=cycle D= day
  Arms: Docetaxel
Drug: Savolitinib — 600 mg QD
  1 cycle = 28 days
  Arms: durvalumab+savolitinib

SUMMARY:
Research Hypothesis Lung cancer is the leading cause of cancer-related mortality in France and in western countries, accounting for more than 1.8 million new cases and 1.5 million deaths worldwide in 2012. Recent advances in the management of patients with Non-small Cell Lung Cancer Patients (NSCLC) include the use of therapies targeting oncogenes but a molecular alteration is currently found in only the half of the non-squamous NSCLC . More recently, immune check point inhibitors (ICI), firstly targeting PD-(L)1, became available and demonstrate an overall survival advantage over standard second-line chemotherapy both in squamous and non-squamous NSCLC. Unfortunately, this global overall survival benefit is driven by approximately 20% of the patient's population while a large majority of patients is in fact progressing in the first weeks of treatment.

In the context of personalized medicine, innovative immunotherapy strategies in oncology are based on the principle of immune-contexture and require:

* The identification of biomarkers for assessing the specific immune-contexture of each patient (microenvironment, tumors and effector cells)
* The development of new treatments targeting their appropriate effector cells in monotherapy or combination treatments.

The current PIONEER-Clinical study is aimed at assessing how to overcome resistance to ICIs monotherapies or ICI in combination with platinum-based chemotherapies, with experimental precision immunotherapies combined to Durvalumab in 2nd, 3rd or 4th line, in advanced NSCLC progressors patients after up to 18more than 6 w. of anti PD (L) 1. for ICIs monotherapies and after more than 12w. of anti PD(L)1 in combination with chemotherapies.

Some supplementary blood and tissue samples are aimed at identification of personalized patients' biomarkers, correlation of them with the efficacy endpoints, in order to better understand mechanisms of resistance and improve their future treatment.

DETAILED DESCRIPTION:
Study Design:

During a mandatory post treatment 28-day wash-out period, 135 advanced NSCLC patients with progressive disease evaluated between 6 and 18w. of a second or third line ICI monotherapy; will undergo a screening visit. After signing an informed written consent, if they are found eligible, their participation in the study will ensue.

Treatment allocation will be performed using the randomization module of the eCRF, :

* Arm A: combination of Durvalumab (MEDI4736) + Monalizumab (IPH2201), to target a PD-L1 co-inhibitory pathway
* Arm B: combination of Durvalumab + oleclumab (MEDI9447), to target limitations of antitumor T-cell immunity caused by adenosine receptor signaling (inclusions closed on May 10, 2021)
* Arm C: combination of Durvalumab + AZD6738, to potentially enhance anti- tumour T-cell responses
* Arm D: a standard third or forth-line chemotherapy maintenance (Docetaxel)
* Arm E : combination of Durvalumab + MET kinase inhibitor Savolitinib (AZD6094)

A maximum of 120 patients will be randomized, with 30 patients per arm (4 arms).

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give a signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent obtained from the patient prior to performing any protocol-related procedures, including screening evaluations.
* Age > 18 years.
* Patients must have histologically confirmed diagnosis of advanced (proven advanced stage) or recurrent NSCLC, (both squamous and non-squamous pathologies are accepted; patients with a mixed NSCLC and SCLC component are ineligible)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Body weight >35kg
* Patients with evidence of radiological progression after more than 6 weeks of a registered second or third line PD1 or PD-L1 inhibitor in monotherapy (to include , Nivolumab, Pembrolizumab, Atezolizumab) or more than 12 weeks for a first line PD-1 or PD-L1 inhibitor in combination with platinum-based chemotherapy.Patients who have received immunotherapy in the maintenance setting can only have had one prior regimen containing PD-1/L1 inhibitor. No intervening treatment between the immunotherapy and entry into this study is permitted.
* Patients with known actionable molecular alteration (EGFR activating mutation, ALK rearrangement, ROS1 rearrangement) should have received a commercially available specific inhibitor
* Patients must have an available archived tissue from a standard tumor biopsy for PD-L1 assessment, done before PD-1 ICI initiation.
* As of Week 1 Day 1, subjects with central nervous system (CNS) metastases must have been treated and must be asymptomatic and meet the following:

  1. No concurrent treatment, inclusive of but not limited to surgery, radiation, and/or corticosteroids
  2. At least 14 days after CNS treatment, clinically stable with no symptoms of CNS metastasis or sequelae of radiation and at least 14 days since last dose of corticosteroids NOTE: Subjects with clinical symptoms or cord compression or with leptomeningeal disease are excluded from the study
* Adequate organ and bone marrow function as defined below:

  1. Haemoglobin ≥10.0 g/dL (transfusion to achieve this level is not permitted within 2 weeks of first study drug administration)
  2. Absolute neutrophil count (ANC) 1.5 x (> 1500 per mm3) (stable off any growth factor within 4 weeks of first study drug administration)
  3. Platelet count ≥100 x 109/L (>100,000 per mm3) (transfusion to achieve this level is not permitted within 2 weeks of first study drug administration)
  4. Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (no upper limit for those patients with persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology, ≤3 x ULN for patients with liver metastases), who will be allowed only in consultation with their physician.
  5. Normal thyroid function, subclinical hypothyroidism (TSH < 10 mIU/mL) or have controlled thyroid disorder
  6. AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
  7. Measured creatinine clearance (CL) >45 mL/min or Calculated creatinine CL>45 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance.
* Women must not be breastfeeding

Exclusion Criteria:

* Individuals deprived of liberty or placed under the authority of a tutor
* Patient unable to understand, read and/or sign an informed consent
* Absence of a measurable target lesion according to RECIST criteria 1.1
* Any symptomatic or untreated brain metastasis
* Any previous treatment with Docetaxel
* Prior randomisation or treatment with durvalumab AZD6738, Medi9447, Monalizumab
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Any previous treatment with a PD1 or PD-L1 inhibitor with the following events:

  1. Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
  2. All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.
  3. Must not have experienced a ≥Grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy.
  4. Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day
  5. No systemic intervening treatment between progression on ICI and entry into this study
* Last dose of immunotherapy ≤21 days prior to the first dose of study drug.
* The patient can receive a stable dose of bisphosphonates or denosumab for bone metastases, before and during the study as long as these were started at least 5 days prior to the study treatment.
* Current or prior use of steroids or other immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which do not exceed 10 mg/day of prednisone, or an equivalent corticosteroid. - Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
* Palliative radiotherapy (to a non target lesion) must have been completed at least 7 days before Cycle 1 Day 1 (with the exception of patients receiving radiation to more than 30% of the bone marrow or with a wide field of radiation who must have completed treatment within 28 days of the first dose of study treatment).
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IMP : patients must have recovered from any effects of any major surgery Note: Localsurgery and other procedures (radiotherapy) of isolated lesions for palliative intent is acceptable.
* History of allogenic organ or stem cell transplantation.
* Active or prior documented autoimmune related inflammatory disorders treated with systemic immunosuppressive drugs within the last 3 months or history of clinically severe auto-immune disease (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]).
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
* Any other malignancy which has been active or treated within the past three years,with the exception of :

  1. cervical intra-epithelial neoplasia,
  2. non-melanoma skin cancer, or lentigo maligna without evidence of disease
  3. ductal Carcinoma in Situ (DCIS),
  4. stage 1 grade 1 endometrial carcinoma,
  5. or other solid tumours curatively treated with no evidence of disease for ≥ 5 years prior to study entry
* History of leptomeningeal carcinomatosis
* Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart) For durvalumab in combination with an agent with pro-arrhythmic potential or where effect of the combination on QT is not known if this criterion should be retained. Patient safety and the cardiac EKG should be consulted as needed.
* History of active primary immunodeficiency
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Receipt of live attenuated vaccine within 30 days prior to the first dose of Investigational Medicinal Product (IMP).

Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.

* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab in combination with an other agent.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.
* A diagnosis of ataxia telangiectasia
* Refractory nausea and vomiting, chronic gastrointestinal diseases or previous significant bowel resection, with clinically significant sequelae
* Patients receiving, or having received, concomitant medications, herbal supplements and/or foods that significantly modulate cytochrome P450 3A4 (CYP3A4) or P-glycoprotein (P-gp) activity (washout periods of 5 half-lives( minimum2 weeks), but 3 weeks for St. John's Wort). NOTE these include common azole antifungals, macrolide antibiotics and other medications.
* Patient has had prescription or non-prescription drugs or other products known to be CYP3A4 and/or CYP2B6 substrates or CYP3A4 and/or CYP2B6 substrates with a narrow therapeutic index. Exposure of other drugs metabolised by CYP3A4 and/or CYP2B6 may be reduced and additional monitoring may be required, see Appendix E.
* The use of herbal supplements or 'folk remedies' (and medications and foods that significantly modulate CYP3A activity) should be discouraged. If deemed necessary, such products may be administered with caution and the reason for use documented in the CRF. Please see Appendix E, for further details.
* Patients with relative hypotension (<90/60 mmHg) or clinically relevant orthostatic hypotension, including a fall in blood pressure of >20 mmHg at screening.
* Any of the following cardiac criteria currently or within the last 6 months (by New York Heart Association (NYHA) ≥ Class 2 where applicable)

  1. Patients at risk of brain perfusion problems, e.g., medical history of carotid stenosis or pre-syncopal or syncopal episodes, history of TIAs
  2. Uncontrolled hypertension (grade 2 or above) requiring clinical intervention
  3. Mean resting corrected QT interval (QTc) >470 msec for females and >450 for men,obtained from 3 electrocardiograms (ECGs) 5-10 minutes apart using the Fredericia formula
  4. Conduction abnormality not controlled with pacemaker or medication e.g. complete left bundle branch block, third degree heart block
  5. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as hypokalaemia, congenital long QT syndrome, immediate family history of long QT syndrome or unexplained sudden death under 40 years of age
  6. Unstable angina pectoris or acute myocardial infarction
  7. Congestive heart failure or known reduced LCEF < 55%
  8. INR ≥1.5 or other evidence of impaired hepatic function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
the 12-week Disease Control Rate | 12 weeks
  in each arm of treatment

SECONDARY OUTCOMES:
Overall Response Rate | 12 months
  the proportion of patients with complete response (CR) or partial response (PR) as best overall response over the treatment period.
Progression-free survival (PFS) | 12 months
PFS Ratio | 12 months
  the date of randomization until the date of event defined as the first documented progression or death from any cause.
Overall Survival (OS) | 6 months
  measured from the date of randomization to the date of death from any cause
Duration of Response | 4years
  measured in to patients whose Best overall response is either CR or PR. It will be measured from the time of first documented response (CR or PR) until the first documented disease progression or death due to underlying cancer.

CONTACTS AND LOCATIONS:
Overall Officials: jean-olivier ARNAUD, Study Director — Assistance Publique -hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France